CLINICAL TRIAL: NCT00570050
Title: A Randomized, Double-blind, Placebo-controlled Cross-over Trial Evaluating the Effect of Intranasal Insulin on Depressive Symptoms in Individuals With Major Depressive Disorder Insufficiently Responsive to Antidepressant Therapy
Brief Title: Effect of Intranasal Insulin on Depressive Symptoms in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Insulin-MDD
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder, Memory, Executive function
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Insulin nasal spray (Experimental)
  Interventions: Drug: Diluent / Insulin; Drug: Insulin / Diluent
- Placebo nasal spray (i.e., no active treatment) (Experimental)
  Interventions: Drug: Diluent / Insulin; Drug: Insulin / Diluent

INTERVENTIONS:
Drug: Diluent / Insulin — Diluent (4 Weeks ) / Intranasal insulin (4 weeks)
Drug: Insulin / Diluent — Intranasal Insulin (4 Weeks ) / Diluent (4 Weeks)

SUMMARY:
The primary aim of the study is to determine whether adjunctive intranasal insulin will exert an antidepressant effect when compared to placebo in adults with major depressive disorder (MDD), insufficiently responsive conventional antidepressants. There are three secondary aims of the study (1) to determine whether adjunctive intranasal insulin will alter emotional processing (i.e., cognitive-affective interface); (2) to determine whether early changes in emotional processing (i.e., after a single dose at 40IU intranasal insulin) predicts symptomatic improvement at study endpoint; and (3) to determine the effect of intranasal insulin on neurocognitive performance (e.g., learning and memory). This initiative represents a proof-of-concept study that insulin is important to depressive symptoms, neurocognitive functioning, and emotional processing deficits in MDD, representing a novel and safe therapeutic avenue.

DETAILED DESCRIPTION:
Emerging evidence for impairments at the cognitive-affective interface, frequently defined as affective cognition, are increasingly being recognized as a core feature of mood disorders, particularly MDD. Individuals with MDD consistently exhibit abnormalities in verbal memory with particular difficulty in memory tasks such as list learning and free recall. The administration of intranasal insulin has been reported to improve verbal memory, declarative memory in individuals with Alzheimer's disease or Mild Cognitive Impairment as well as measures of mood (e.g., overall feeling of well-being, self-esteem, and depression) in healthy volunteers. The effect of intranasal insulin on any measure of neurocognitive function and emotional processing in MDD is currently unknown.

Thirty participants between the ages of 18 and 60 with DSM-IV-TR defined MDD [confirmed by the Mini International Neuropsychiatric Interview (MINI)] will be enrolled. Individuals below the age of 18 and over 60 are excluded as they are not seen at the recruiting center. Enrollment into the study is voluntary. Eligible participants will provide written informed consent. Participants will be enrolled from the outpatient Mood Disorders Psychopharmacology Unit (MDPU), University Health Network (UHN), University of Toronto.

The MDPU case report form will gather information on the participant's course of illness variables. Conventional pharmacological treatments for MDD will be permitted (e.g., conventional antidepressants). Conventional unimodal antidepressants modulate cerebral glucose metabolism; as such, they will be kept consistent throughout the duration of the study and will not be altered from the point of randomization to study endpoint. Antidepressants and augmentation strategies with significant anti-cholinergic potential (e.g., paroxetine, tricyclic antidepressants) as well as benzodiazepines will be exclusionary as they may negatively affect neurocognitive function.

Participants will be excluded if they are receiving corticosteroids or antihypertensive medications; misused substance or alcohol in the past 3 months; received electroconvulsive therapy in the last 1 year; or have a neurological or medically unstable condition. Another exclusion criterion includes the inability to provide written informed consent. The Montgomery-Asberg Depression Rating Scale (MADRS) and Hamilton Depression Rating Scale 17-Item (HAM-D-17) will be administered at baseline and weekly throughout the 8 weeks of treatment assignment. Participants who are actively suicidal or evaluated as being a suicide risk will also be excluded. Other reasons for discontinuation are impaired fasting glucose (i.e., 6.1 - 6.9 mmol/L), and non-compliance (i.e., failure to administer ≥ 80% of the assigned treatment in any week).

The ongoing provision of care is not contingent on enrollment and/or completion of the study protocol. Furthermore, there will be ongoing communication with the participant's primary care provider in regards to their participation in this study.

This is a randomized double-blind, placebo-controlled, cross-over study. The initial visit entails the provision of detailed study information to the patient and obtainment of written informed consent from the participant. The participant will then meet a research team member at a later date for a screening visit. This study requires a total of 12 visits.

Full neuropsychological testing will be conducted at 4 time points:

1. Baseline1 (Visit 3)
2. Endpoint1 (Visit 7)
3. Baseline2 (Visit 8)
4. Endpoint2 (Visit 12)

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder - current depression

Exclusion Criteria:

* Unstable medical conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 9 weeks
  Score form baseline to end of each treatment phase.

SECONDARY OUTCOMES:
Affective Go/No-Go and Emotional Recognition Tasks; CGI Severity of Illness, Improvements in subjective mood (PANAS) and quality of life (Q-LES-Q) | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roger S McIntyre, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada